CLINICAL TRIAL: NCT01259622
Title: A mulTi-center, Randomized, doUble-bliNded, Placebo-controlled Dose-escalating Study of the Effects of K201 on the RestorAtion of Sinus Rhythm in Subjects With Symptomatic Atrial Fibrillation of Recent Onset
Brief Title: Effects of Intravenous K201 on the Restoration of Sinus Rhythm in Subjects With Symptomatic Atrial Fibrillation
Acronym: TUNDRA-AF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sequel Pharmaceuticals, Inc (Industry)
Responsible Party: Howard C Dittrich, MD, Sequel Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJI-202
Record Dates: First submitted 2010-12-12; First posted 2010-12-14 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sodium Chloride; K201 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: saline
- K201 (Experimental): intravenous K201
  Interventions: Drug: K201

INTERVENTIONS:
Drug: saline — intravenous infusion
  Arms: placebo
Drug: K201 — intravenous infusion
  Arms: K201

SUMMARY:
The purpose of this study is to evaluate the effects of a single intravenous infusion of K201 compared to placebo in a dose escalating manner on conversion to sinus rhythm, reduction of subject's symptom score, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial fibrillation for more than 3 hours and less than 7 days (as dated by symptoms).
* Atrial fibrillation documented by ECG at the start of study drug infusion.

Exclusion Criteria:

* Previous exposure to K201
* QTcF (Fridericia correction) >440 ms
* QRS interval > 140 ms
* Paced atrial or paced ventricular rhythm on ECG
* History of receiving another intravenous Class I or Class III antiarrhythmic drug within 3 days of randomization
* History of amiodarone (oral or IV) in the last 3 months.
* Clinical evidence or history of acute coronary syndrome (e.g. myocardial infarction, unstable angina) within 30 days prior to randomization
* History of failed electrical cardioversion at any time in the past
* History of polymorphic ventricular tachycardia (e.g. torsades des pointes)
* History or family history of Long QT Syndrome
* History of ventricular tachycardia requiring drug or device therapy
* Ejection fraction of 40% or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects who convert to sinus rhythm | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chamberlin, MD, Study Director — Sequel Pharmaceuticals
Locations (17):
- Denmark (14):
  - Copenhagen
  - Esbjerg
  - Glostrup Municipality
  - Haderslev
  - Hellerup
  - Herlev
  - Hvidovre
  - Kolding
  - Odense
  - Roskilde
  - Silkeborg
  - Svendborg
  - Varde
  - Viborg
- Israel (3):
  - Ashkelon
  - Rehovot
  - Safed